CLINICAL TRIAL: NCT01751776
Title: A Randomised, Double-blind, Placebo-controlled Trial for Establishing Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Clinical Efficacy of Multiple Subcutaneous Doses of BI 655064 in Healthy Volunteers and in Rheumatoid Arthritis Patients With Prior Inadequate Response to Methotrexate Therapy
Brief Title: Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Clinical Effects of Multiple Rising Subcutaneous Doses of BI 655064 in Healthy Volunteers and in Rheumatoid Arthritis Patients With Prior Inadequate Response to Methotrexate Therapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1293.2; 2012-004090-16 (EudraCT Number: EudraCT)
Record Dates: First submitted 2012-12-14; First posted 2012-12-18 (Estimated); Results first posted 2024-03-21 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2023-09

CONDITIONS: Arthritis, Rheumatoid; Healthy
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — BI 655064

ARMS (8):
- Part 1, Placebo BI 655064 80/120mg (HV) (Placebo Comparator): Part 1, Healthy volunteers (HV): Placebo matching BI 655064 80 or 120 milligram (mg) injected subcutaneous on days 1, 8, 15, and 22 (once weekly, for 4 weeks) followed by 6 weeks follow-up period.
  Interventions: Drug: Placebo matching BI 655064
- Part 1, Placebo BI 655064 180/240mg (HV) (Placebo Comparator): Part 1, Healthy volunteers (HV): Placebo matching BI 655064 180 or 240 mg injected subcutaneous on days 1, 8, 15, and 22 (once weekly, for 4 weeks) followed by 6 weeks (180mg dosing group) or 8 weeks (240mg dosing group) follow-up period.
  Interventions: Drug: Placebo matching BI 655064
- Part 1, BI 655064 80mg (HV) (Experimental): Part 1, Healthy volunteers (HV): 80 mg of BI 655064 injected subcutaneous on days 1, 8, 15, and 22 (once weekly, for 4 weeks) followed by 6 weeks follow-up period.
  Interventions: Drug: BI 655064
- Part 1, BI 655064 120mg (HV) (Experimental): Part 1, Healthy volunteers (HV): 120 mg of BI 655064 injected subcutaneous on days 1, 8, 15, and 22 (once weekly, for 4 weeks) followed by 6 weeks follow-up period.
  Interventions: Drug: BI 655064
- Part 1, BI 655064 180mg (HV) (Experimental): Part 1, Healthy volunteers (HV): 180 mg of BI 655064 injected subcutaneous on days 1, 8, 15, and 22 (once weekly, for 4 weeks) followed by 6 weeks follow-up period.
  Interventions: Drug: BI 655064
- Part 1, BI 655064 240mg (HV) (Experimental): Part 1, Healthy volunteers (HV): 240mg of BI 655064 injected subcutaneous on days 1, 8, 15, and 22 (once weekly, for 4 weeks) followed by 8 weeks follow-up period.
  Interventions: Drug: BI 655064
- Part 2, Placebo BI 655064 120mg (RA) (Placebo Comparator): Part 2, patients with Rheumatoid arthritis (RA) who had prior inadequate response to Methotrexat (MTX) therapy: Placebo matching BI 655064 120 milligram (mg) injected subcutaneous on days 1, 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, and 78 (once weekly for 12 weeks) followed by 8 weeks follow-up period.
  Interventions: Drug: Placebo matching BI 655064
- Part 2, BI 655064 120mg (RA) (Experimental): Part 2, patients with RA who had prior inadequate response to MTX therapy: 120 milligram (mg) of BI 655064 injected subcutaneous on days 1, 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, and 78 (once weekly for 12 weeks) followed by 8 weeks follow-up period.
  Interventions: Drug: BI 655064

INTERVENTIONS:
Drug: Placebo matching BI 655064 — Placebo matching BI 655064 injected subcutaneous.
  Arms: Part 1, Placebo BI 655064 180/240mg (HV); Part 1, Placebo BI 655064 80/120mg (HV); Part 2, Placebo BI 655064 120mg (RA)
Drug: BI 655064 — BI 655064 injected subcutaneous
  Arms: Part 1, BI 655064 120mg (HV); Part 1, BI 655064 180mg (HV); Part 1, BI 655064 240mg (HV); Part 1, BI 655064 80mg (HV); Part 2, BI 655064 120mg (RA)

SUMMARY:
To evaluate the safety and tolerability of multiple doses of BI 655064 administered subcutaneously in healthy volunteers (HVs) and in rheumatoid arthritis (RA) patients. To explore the pharmacokinetic (PK) and pharmacodynamic (PD) parameters of multiple doses of BI 655064 in healthy volunteers (HVs) and rheumatoid arthritis (RA) patients. To assess clinical effect of BI 655064 in RA patients with prior inadequate response to methotrexate (MTX) after 12 weeks of treatment

ELIGIBILITY:
Inclusion criteria:

Part 1 (phase Ib) (HVs):

1. Healthy males and females according to the investigators assessment, as based on the following criteria: a complete medical history including a physical examination, vital signs (BP, PR), 12-lead ECG, and clinical laboratory tests
2. Age >= 18 and <= 60 years
3. Body Mass Index >= 18.5 and <= 29.9 kg/m2
4. Signed and dated written informed consent prior to admission to the study in accordance with GCP and the local legislation
5. Female subjects who meet any of the following criteria from at least 30 days before the first study drug administration and until 30 days after trial completion:

   * using adequate contraception, e.g. any of the following methods plus condom: implants, injectables, combined oral contraceptives, intrauterine device (IUD)
   * sexually abstinent
   * have a vasectomised sexual partner (vasectomy at least 1 year prior to enrolment)
   * surgically sterilised (including hysterectomy)
   * postmenopausal defined as at least 1 year of spontaneous amenorrhea (in questionable cases a blood sample with simultaneous levels of follicle stimulating hormone (FSH) above 40 U/L and estradiol below 30 ng/L is confirmatory)

Part 2 (phase IIa) (RA Patients):

1. Age >= 18 and <= 70 years
2. Patients classified as having RA according to the 1987 ACR Classification Criteria
3. Inadequate clinical response to methotrexate monotherapy defined as moderate/high active disease after oral or s.c. MTX treatment given continuously for at least 3 months and for the last 6 weeks before screening at a stable weekly dose >=15mg. For patients who do not tolerate the minimum weekly dose of at least 15 mg due to side effects, a stable weekly dose as low as 7.5 mg is also permitted.
4. DAS28 4v-CRP >= 3.5 with >= 6 tender and >= 6 swollen joints out of 68/66 joint count at screening and confirmed by >= 6 tender and >= 6 swollen joints out of 68/66 joint count only at randomisation visit (Visit 2)
5. Serum CRP level >= 0.8 mg/dL or ESR >= 28 mm/1h at screening
6. Anti-CCP2 or Rheumatoid Factor positivity as per the limits of used assay at screening
7. Female patients who meet any of the following criteria from at least 30 days before the first study drug administration and until at least 6 months after last dose of MTX taken in the current trial:

   using adequate contraception, e.g. any of the following methods plus condom: implants, injectables, combined oral contraceptives, intrauterine device (IUD)
   * sexually abstinent
   * have a vasectomised sexual partner (vasectomy at least 1 year prior to enrolment)
   * surgically sterilised (including hysterectomy)
   * postmenopausal defined as at least 1 year of spontaneous amenorrhea (in questionable cases a blood sample with simultaneous levels of follicle stimulating hormone (FSH) above 40 U/L and estradiol below 30 ng/L is confirmatory)

   OR

   Male patients who:
   * are documented to be sterile or consistently and correctly use a condom while their female partners (if of childbearing potential) agree to use any of the following adequate contraception methods: implants, injectables, combined oral contraceptives, intrauterine device (IUD) from the date of screening until at least 6 months after the last dose of MTX taken in the current trial
   * don¿t donate any sperm sample for procreation purposes, from the date of screening until at least 6 months after last dose of MTX taken in the current trial.
8. Signed and dated written informed consent prior to admission to the study in accordance with GCP and local legislation

Exclusion criteria:

Part 1 (phase Ib in HVs):

1. Any finding in the medical examination (including BP, PR or ECG) deviating from normal and judged clinically relevant by the investigator
2. Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
3. Any evidence of a concomitant disease judged clinically relevant by the investigator
4. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
5. Diseases of the central nervous system (such as epilepsy), other neurological disorders or psychiatric disorders
6. History of relevant orthostatic hypotension, fainting spells, or blackouts
7. History of relevant allergy/hypersensitivity (including allergy to the trial medication or its excipients)

9. Within 10 days prior to administration of trial medication, use of drugs that might reasonably influence the results of the trial 12. Alcohol abuse (consumption of more than 140 g/week in females and 210 g/week in males) 13. Drug abuse or positive drug screen 17. Chronic or relevant acute infections, including but not limited to HIV, Hepatitis B and C and tuberculosis (including a history of clinical TB and/or a positive QuantiFERON TB-Gold test) 18. Subject is assessed by the investigator as unsuitable for inclusion e.g. considered not able to understand and comply with study requirements or has a condition that would not allow safe participation in the study 19. Positive pregnancy test, pregnancy or plans to become pregnant within 30 days after study completion 20. Lactation

Further exclusion criteria applicable for part 1 only are given in the CTP.

Part 2 (phase IIa in RA patients):

Part 1 (phase Ib) exclusion criteria 7, 9, 12, 13 and 17-20 plus:

1. Current or previous use of more than two anti-TNF biologic drugs or use of other biologic agent targeting any other approved mechanism (any biologic drug with mechanism of action other than direct anti-TNF blockade, (e.g. CTLA4, anti-IL6, or anti CD-20) or new oral compounds targeting any other approved mechanism (e.g. JAK inhibitors) for treating RA.
2. Current or previous participation in a clinical trial testing an investigational drug for RA within 3 months prior to screening or within 5 half-lives of the investigational drug, whichever is longer , except of previous participation in trials testing NSAIDs, corticosteroids, analgesics or patients documented as receiving placebo in previous RA trials.
3. DAS28 < 3.2 in at least 2 occasions during the last 6 months before screening
4. RA patients with severe disability (functional class IV) or with confirmed severe systemic manifestations e.g. known amyloidosis, Felty´s syndrome, lymphoproliferative disorders, rheumatoid vasculitis
5. Treatment with any standard DMARD except MTX (including but not limited to sulfasalazine, leflunomide, hydroxychloroquine, D-penicillamine
6. Impaired hepatic function, defined as serum AST/ALT, bilirubin or alkaline phosphatase levels > 2 x ULN
7. Impaired renal function defined as calculated creatinine clearance < 50ml/min
8. Pre-existing blood dyscrasias e.g. bone marrow hypoplasia, significant anaemia, leucopenia or thrombocytopenia
9. Hypersensitivity to MTX or any of its excipients
10. Previous intolerance to MTX as the main cause for stopping treatment (instead of lack of efficacy)
11. Any active or suspected malignancy or history of documented malignancy within the last 5 years before screening, except appropriately treated basal cell carcinoma of the skin or in situ carcinoma of uterine cervix.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2012-12-18 (Actual); Primary Completion 2015-03-02 (Actual); Study Completion 2015-04-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (25):
- Czechia (3):
  - 1293.2.00049 Boehringer Ingelheim Investigational Site, Olomouc
  - 1293.2.00024 Boehringer Ingelheim Investigational Site, Uherské Hradiště
  - 1293.2.00028 Boehringer Ingelheim Investigational Site, Zlín
- Germany (5):
  - 1293.2.00015 Boehringer Ingelheim Investigational Site, Bad Kreuznach
  - 1293.2.00010 Boehringer Ingelheim Investigational Site, Berlin
  - 1293.2.00013 Boehringer Ingelheim Investigational Site, Berlin
  - 1293.2.00043 Boehringer Ingelheim Investigational Site, München
  - 1293.2.00012 Boehringer Ingelheim Investigational Site, Zerbst
- Netherlands (4):
  - 1293.2.00031 Boehringer Ingelheim Investigational Site, Amsterdam
  - 1293.2.00032 Boehringer Ingelheim Investigational Site, Leeuwarden
  - 1293.2.00038 Boehringer Ingelheim Investigational Site, Leiden
  - 1293.2.00040 Boehringer Ingelheim Investigational Site, Sneek
- 1293.2.00001 Boehringer Ingelheim Investigational Site, Grafton Auckland NZ, New Zealand
- Poland (7):
  - 1293.2.00039 Boehringer Ingelheim Investigational Site, Bialystok
  - 1293.2.00034 Boehringer Ingelheim Investigational Site, Bydgoszcz
  - 1293.2.00041 Boehringer Ingelheim Investigational Site, Bydgoszcz
  - 1293.2.00025 Boehringer Ingelheim Investigational Site, Lublin
  - 1293.2.00050 Boehringer Ingelheim Investigational Site, Poznan
  - 1293.2.00023 Boehringer Ingelheim Investigational Site, Warsaw
  - 1293.2.00026 Boehringer Ingelheim Investigational Site, Warsaw
- Spain (5):
  - 1293.2.00021 Boehringer Ingelheim Investigational Site, A Coruña
  - 1293.2.00017 Boehringer Ingelheim Investigational Site, Barcelona
  - 1293.2.00022 Boehringer Ingelheim Investigational Site, Granada
  - 1293.2.00016 Boehringer Ingelheim Investigational Site, La Laguna (Sta Cruz Tenerife)
  - 1293.2.00020 Boehringer Ingelheim Investigational Site, Santiago de Compostela

REFERENCES:
- [Derived] Visvanathan S, Daniluk S, Ptaszynski R, Muller-Ladner U, Ramanujam M, Rosenstock B, Eleftheraki AG, Vinisko R, Petrikova A, Kellner H, Dokoupilova E, Kwiatkowska B, Alten R, Schwabe C, Baum P, Joseph D, Fine JS, Padula SJ, Steffgen J. Effects of BI 655064, an antagonistic anti-CD40 antibody, on clinical and biomarker variables in patients with active rheumatoid arthritis: a randomised, double-blind, placebo-controlled, phase IIa study. Ann Rheum Dis. 2019 Jun;78(6):754-760. doi: 10.1136/annrheumdis-2018-214729. Epub 2019 Mar 22. PMID 30902820

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Part 1 (Phase Ib multiple rising dose): 40 healthy volunteers were recruited, in 4 sequential groups of 10 subjects (8 of them received active drug, 2 placebo) each. Thereafter, part 2 (Phase 2a): 67 patients with Rheumatoid Arthritis(RA), who had prior inadequate response to Methotrexate (MTX)treatment, were randomised into 2 arms.
Pre-assignment Details: All subjects were screened for eligibility to participate in trial. Subjects attended specialist sites to ensure that they (the subjects) met all implemented inclusion/exclusion criteria. Subjects were not to be randomised to trial drug if any of the specific entry criteria was violated.
Period: Overall Study
Arm/Group | Part 1, Placebo BI 655064 80/120mg (HV) | Part 1, Placebo BI 655064 180/240mg (HV) | Part 1, BI 655064 80mg (HV) | Part 1, BI 655064 120mg (HV) | Part 1, BI 655064 180mg (HV) | Part 1, BI 655064 240mg (HV) | Part 2, Placebo BI 655064 120mg (RA) | Part 2, BI 655064 120mg (RA)
Started | 4 | 4 | 8 | 8 | 8 | 8 | 23 | 44
Completed | 4 | 4 | 8 | 8 | 8 | 8 | 19 | 40
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 4
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 2
Not completed — Consent withdrawn | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Other reason not specified above | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Treated set (TS): This patient set includes all subjects who were dispensed study medication and were documented to have taken at least one dose of investigational treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1, Placebo BI 655064 80/120mg (HV) | Part 1, Placebo BI 655064 180/240mg (HV) | Part 1, BI 655064 80mg (HV) | Part 1, BI 655064 120mg (HV) | Part 1, BI 655064 180mg (HV) | Part 1, BI 655064 240mg (HV) | Part 2, Placebo BI 655064 120mg (RA) | Part 2, BI 655064 120mg (RA) | Total
Number analyzed (Participants) | 4 | 4 | 8 | 8 | 8 | 8 | 23 | 44 | 107
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: As pre-specified in the protocol, subjects in part 1 and part 2 were analyzed separately.
  years
    Part 1: number analyzed (Participants) | 4 | 4 | 8 | 8 | 8 | 8 | 0 | 0 | 40
    Part 1 | 21.5 (1.3) | 34.0 (15.4) | 25.9 (4.1) | 31.4 (13.3) | 37.3 (10.8) | 29.5 (10.6) |  |  | 30.4 (10.8)
    Part 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 23 | 44 | 67
    Part 2 |  |  |  |  |  |  | 55.1 (8.3) | 53.7 (13.3) | 54.2 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 2 | 0 | 2 | 1 | 18 | 37 | 62
  Male | 4 | 2 | 6 | 8 | 6 | 7 | 5 | 7 | 45
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 0 | 0 | 3 | 2 | 0 | 0 | 7
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 3 | 2 | 6 | 7 | 5 | 6 | 23 | 43 | 95
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Cmax After the First and Last Dose
Description: Part 1: This outcome measure presents the maximum measured concentration of BI 655064 in plasma (Cmax) after the first and last (fourth) dose. More detailed time frame: Pharmacokinetic (PK) sample times: 0:30 hour (h) prior first administration of BI 655064 and 1 h, 8 h, 12 h, 24 h, 48 h, 72 h, 84 h, 96 h, 108 h, 120 h, 144 h, 167:30 h, 335:30 h, 503:30 h, 505 h, 516 h, 528 h, 552 h, 576 h, 600 h, 624 h, 648 h, 672 h, 696 h, 744 h, 816 h, 912 h, 1008 h, 1176 h, 1344 h, 1512 h, 1848 h thereafter; further administration times for BI 655064: 168 h, 336 h, and 504 h after first administration.
Time Frame: From first day of drug administration till end of trial, up to 77 days. Detailed PK can be found in the endpoint description.
Population: All subjects were treated and and provided data for at least 1 primary pharmacokinetic (PK) endpoint and therefore all subjects were also included in the PK set (PKS).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram (µg)/ millilitre (mL)
Arm/Group | Part 1, BI 655064 80mg (HV) | Part 1, BI 655064 120mg (HV) | Part 1, BI 655064 180mg (HV) | Part 1, BI 655064 240mg (HV)
Number analyzed (Participants) | 8 | 8 | 8 | 8
microgram (µg)/ millilitre (mL)
  after the first dose | 1.59 (492) | 7.70 (29.5) | 9.87 (67.8) | 18.0 (46.3)
  after the last (fourth) dose | 13.1 (59.1) | 28.7 (35.6) | 39.8 (37.4) | 68.4 (21.9)
Statistical Analysis 1: Comparison: Part 1, BI 655064 80mg (HV) vs Part 1, BI 655064 120mg (HV) vs Part 1, BI 655064 180mg (HV) vs Part 1, BI 655064 240mg (HV); Dose proportionality for Cmax was explored after the first adminstration of BI 65564 on Day 1; Test type: Superiority or Other; Slope = 2.0506, 95% CI 2-sided [1.1843 to 2.9168], Standard Error of Mean 0.4242 — Dose proportionality was explored using a regression model. Based on the estimate for the slope parameter, a 2-sided 95% CI was computed. Perfect dose proportionality would correspond to a slope of 1. PK endpoints on the log-transformed scale
Statistical Analysis 2: Comparison: Part 1, BI 655064 80mg (HV) vs Part 1, BI 655064 120mg (HV) vs Part 1, BI 655064 180mg (HV) vs Part 1, BI 655064 240mg (HV); Dose proportionality for Cmax was explored after the last (fourth) adminstration of BI 65564 on Day 22; Test type: Superiority or Other; Slope = 1.4227, 95% CI 2-sided [1.0869 to 1.7584], Standard Error of Mean 0.1644 — [estimate comment as in outcome 1, analysis 1]

2. Primary Outcome: Part 1: AUC 0-infinity After the Last Dose
Description: Part 1: Area under the concentration-time curve of BI 655064 in plasma over the time interval from 0 extrapolated to infinite (AUC 0-infinity).
Time Frame: PK sample times: 1 h, 12 h, 24 h, 48 h, 72 h, 96 h, 120 h, 144 h, 168 h, 192 h, 240 h, 312 h, 408 h, 504 h, 672 h, 840 h, 1008 h, 1344 h after the last administration of BI 655064 on day 22
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg* hours (h)/mL
Arm/Group | Part 1, BI 655064 80mg (HV) | Part 1, BI 655064 120mg (HV) | Part 1, BI 655064 180mg (HV) | Part 1, BI 655064 240mg (HV)
Number analyzed (Participants) | 8 | 8 | 8 | 8
µg* hours (h)/mL | 3940 (53.9) | 11000 (42.5) | 19200 (41.1) | 39300 (26.1)
Statistical Analysis 1: Comparison: Part 1, BI 655064 80mg (HV) vs Part 1, BI 655064 120mg (HV) vs Part 1, BI 655064 180mg (HV) vs Part 1, BI 655064 240mg (HV); Dose proportionality for AUC 0-infinity was explored after the last adminstration of BI 65564 on Day 22; Test type: Superiority or Other; Slope = 2.0091, 95% CI 2-sided [1.6607 to 2.3575], Standard Error of Mean 0.1706 — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: Part 1: AUCtau After the Last Dose
Description: Area under the concentration-time curve of BI 655064 in plasma after the 4th dose over a uniform dosing interval t (AUC t,4) after the first and 4th dose. AUCtau is synonymous with AUC0-168.
Time Frame: PK sample times: 1 h, 12 h, 24 h, 48 h, 72 h, 96 h, 120 h, 144 h, 168 h, 192 h, 240 h, 312 h, 408 h, 504 h, 672 h, 840 h, 1008 h, 1344 h after the last administration of trial drug on day 22
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg*h/mL
Arm/Group | Part 1, BI 655064 80mg (HV) | Part 1, BI 655064 120mg (HV) | Part 1, BI 655064 180mg (HV) | Part 1, BI 655064 240mg (HV)
Number analyzed (Participants) | 8 | 8 | 8 | 8
µg*h/mL | 1790 (56.4) | 4140 (35.4) | 5470 (37.4) | 9460 (22.4)
Statistical Analysis 1: Comparison: Part 1, BI 655064 80mg (HV) vs Part 1, BI 655064 120mg (HV) vs Part 1, BI 655064 180mg (HV) vs Part 1, BI 655064 240mg (HV); Dose proportionality for AUCtau was explored after the last administration of BI 65564 on Day 22; Test type: Superiority or Other; Slope = 1.4225, 95% CI 2-sided [1.0876 to 1.7574], Standard Error of Mean 0.1640 — [estimate comment as in outcome 1, analysis 1]

4. Primary Outcome: Part 1: Percentage of Subjects With Drug Related Adverse Events
Description: In Part 1 (Phase Ib): The primary safety endpoint was the percentage of subjects with AEs related to treatment with trial medication.
Time Frame: from first administration of study medication (day 1) up to day 64 (dosing groups 80, 120, 180mg) or up to day 78 post-treatment (dosing group 240mg)
Population: TS
Measure: Number; unit: Percentage of participants
Groups:
- Part 1, Placebo BI 655064 (HV): Part 1, Healthy volunteers (HV): Placebo of BI 655064 injected subcutaneous on days 1, 8, 15, and 22 (once weekly, for 4 weeks) followed by a 6 weeks (120mg dosing group) or a 8 weeks (240mg dosing group) follow-up period. Within each dose group two subjects were to receive placebo.
Arm/Group | Part 1, Placebo BI 655064 (HV) | Part 1, BI 655064 80mg (HV) | Part 1, BI 655064 120mg (HV) | Part 1, BI 655064 180mg (HV) | Part 1, BI 655064 240mg (HV)
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8
Percentage of participants | 50.0 | 25.0 | 12.5 | 50.0 | 0.0

5. Primary Outcome: Part 2: American College of Rheumatology (ACR)20 Response Rate at Week 12
Description: ACR 20 criteria at week 12 relative to the patient's status at baseline: that is, at least 20 percent (%) improvement in swollen joint count, at least 20% improvement in tender joint count, and at least 20% improvement in ≥3 of the following 5 variables: 1) patient's assessment of pain on the visual analogue scale (VAS), rated on a scale of 1 to 10; 2) patient's global assessment of disease on the VAS, rated on a scale of 1 to 10; 3) investigator's global assessment of disease on the VAS; 4) patient's assessment of disability on the health assessment questionnaire (HAQ), rated on a scale of 1 to 3; and 5) concentrations of acute phase reactants. For all scales (1-4): smaller values better. The ACR20 were evaluated descriptively. The data were analysed with a Bayesian approach using an informative prior for the placebo treatment group; predictive probability that the treatment difference was larger than 0%, 5%, 10%, 15%, 20%, 25%, 30%, 35%, 40% or 45% was to be evaluated.
Time Frame: at week 12 (day 85) from the initiation of study treatment
Population: The full analysis set (FAS) included 66 of 67 randomised and treated patients; 1 patient (placebo group) was excluded due to insufficient efficacy data (excluded due to important protocol violations). Noncompleters were assumed to be failures (NCF).
Measure: Number; unit: Percentage of participants
Groups:
- Part 2, Placebo: Part 2, patients with Rheumatoid arthritis (RA) who had prior inadequate response to Methotrexat (MTX) therapy: Placebo matching to BI 655064 120 milligram (mg) injected subcutaneous on days 1, 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, and 78 (once weekly for 12 weeks) followed by 8 weeks follow-up period.
Arm/Group | Part 2, Placebo | Part 2, BI 655064 120mg (RA)
Number analyzed (Participants) | 22 | 44
Percentage of participants | 45.5 | 68.2
Statistical Analysis 1: Comparison: Part 2, Placebo vs Part 2, BI 655064 120mg (RA); Observed difference of ACR20 response for BI 120mg - Placebo; Test type: Other; Mean Difference (Net) = 22.7 — Mean Difference in percentage
Statistical Analysis 2: Comparison: Part 2, Placebo vs Part 2, BI 655064 120mg (RA); Expected difference of ACR20 response for BI 120mg - Placebo; Test type: Other — Evaluation of the difference in ACR20 response rates using a Bayesian approach. Results based on 1000000 simulations of the posterior distribution; for the treatment group a non-informative beta (0,0) prior was used; for the placebo group, an informative beta (5.5, 16.5) prior was used; prior to any imputation, assessments up to the End of Trial (EoT) visit were mapped to an on-treatment visit window (Visit 4/Week 2 - Visit 14 (EoT)/Week 12) relative to the day of the first dose; Mean Difference (Net) = 33.0 — Mean Difference in percentage
Statistical Analysis 3: Comparison: Part 2, Placebo vs Part 2, BI 655064 120mg (RA); Probability that difference of ACR20 response for BI 120mg - Placebo is larger than 0%; Test type: Other — [test comment as in outcome 5, analysis 2]; Probability in percentage = 99.9
Statistical Analysis 4: Comparison: Part 2, Placebo vs Part 2, BI 655064 120mg (RA); Probability that difference of ACR20 response for BI 120mg - Placebo is larger than 5%; Test type: Other — [test comment as in outcome 5, analysis 2]; Probability in percentage = 99.7
Statistical Analysis 5: Comparison: Part 2, Placebo vs Part 2, BI 655064 120mg (RA); Probability that difference of ACR20 response for BI 120mg - Placebo is larger than 10%; Test type: Other — [test comment as in outcome 5, analysis 2]; Probability in percentage = 98.7
Statistical Analysis 6: Comparison: Part 2, Placebo vs Part 2, BI 655064 120mg (RA); Probability that difference of ACR20 response for BI 120mg - Placebo is larger than 15%; Test type: Other — [test comment as in outcome 5, analysis 2]; Probability in percentage = 96.0
Statistical Analysis 7: Comparison: Part 2, Placebo vs Part 2, BI 655064 120mg (RA); Probability that difference of ACR20 response for BI 120mg - Placebo is larger than 20%; Test type: Other — [test comment as in outcome 5, analysis 2]; Probability in percentage = 90.0
Statistical Analysis 8: Comparison: Part 2, Placebo vs Part 2, BI 655064 120mg (RA); Probability that difference of ACR20 response for BI 120mg - Placebo is larger than 25%; Test type: Other — [test comment as in outcome 5, analysis 2]; Probability in percentage = 79.0
Statistical Analysis 9: Comparison: Part 2, Placebo vs Part 2, BI 655064 120mg (RA); Probability that difference of ACR20 response for BI 120mg - Placebo is larger than 30%; Test type: Other — [test comment as in outcome 5, analysis 2]; Probability in percentage = 62.5
Statistical Analysis 10: Comparison: Part 2, Placebo vs Part 2, BI 655064 120mg (RA); Probability that difference of ACR20 response for BI 120mg - Placebo is larger than 35%; Test type: Other — [test comment as in outcome 5, analysis 2]; Probability in percentage = 42.9
Statistical Analysis 11: Comparison: Part 2, Placebo vs Part 2, BI 655064 120mg (RA); Probability that difference of ACR20 response for BI 120mg - Placebo is larger than 40%; Test type: Other — [test comment as in outcome 5, analysis 2]; Probability in percentage = 24.5
Statistical Analysis 12: Comparison: Part 2, Placebo vs Part 2, BI 655064 120mg (RA); Probability that difference of ACR20 response for BI 120mg - Placebo is larger than 45%; Test type: Other — [test comment as in outcome 5, analysis 2]; Probability in percentage = 11.1

6. Secondary Outcome: Part 2: ACR50 Response Rates at Week 12
Description: ACR 50 criteria at week 12 relative to the patient's status at baseline: that is, at least 50 % improvement in swollen joint count, at least 50% improvement in tender joint count, and at least 50% improvement in ≥3 of the following 5 variables: 1) patient's assessment of pain on the visual analogue scale (VAS), rated on a scale of 1 to 10; 2) patient's global assessment of disease on the VAS, rated on a scale of 1 to 10; 3) investigator's global assessment of disease on the VAS; 4) patient's assessment of disability on the health assessment questionnaire (HAQ), rated on a scale of 1 to 3; and 5) concentrations of acute phase reactants. For all scales (1-4): smaller values better. The percentage of subjects with ACR50 response is presented.
Time Frame: at week 12 (day 85)
Population: FAS (NCF)
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part 2, Placebo | Part 2, BI 655064 120mg (RA)
Number analyzed (Participants) | 22 | 44
Percentage of participants
  unadjusted | 18.2 [5.2 to 40.3] | 36.4 [22.4 to 52.2]
  adjusted | 15.6 [5.5 to 36.9] | 35.6 [22.3 to 51.5]
Statistical Analysis 1: Comparison: Part 2, Placebo vs Part 2, BI 655064 120mg (RA); unadjusted; Test type: Superiority or Other; p = 0.0754, One-sided exact test (see description); One-sided exact test for superiority testing; Risk difference, unadjusted = 18.2, 95% CI 2-sided [-6.6 to 38.6] — The exact 95% confidence interval was calculated by Clopper and Pearson
Statistical Analysis 2: Comparison: Part 2, Placebo vs Part 2, BI 655064 120mg (RA); adjusted; Test type: Superiority or Other; risk difference, adjusted = 20.0, 95% CI 2-sided [-4.6 to 39.0] — The 95 % confidence interval was determined by root method to determine the cumulative distribution function. Adjusted for treatment, region and anti-Tumour Necrosis Factor (TNF)

7. Secondary Outcome: Part 2: ACR70 Response Rates at Week 12
Description: ACR70 criteria at week 12 relative to the patient's status at baseline: that is, at least 70 % improvement in swollen joint count, at least 70% improvement in tender joint count, and at least 70% improvement in ≥3 of the following 5 variables: 1) patient's assessment of pain on the visual analogue scale (VAS), rated on a scale of 1 to 10; 2) patient's global assessment of disease on the VAS, rated on a scale of 1 to 10; 3) investigator's global assessment of disease on the VAS; 4) patient's assessment of disability on the health assessment questionnaire (HAQ), rated on a scale of 1 to 3; and 5) concentrations of acute phase reactants. For all scales (1-4): smaller values better). The percentage of subjects with ACR50 response is presented.
Time Frame: at week 12 (day 85)
Population: FAS (NCF)
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part 2, Placebo | Part 2, BI 655064 120mg (RA)
Number analyzed (Participants) | 22 | 44
Percentage of participants
  unadjusted | 13.6 [2.9 to 34.9] | 18.2 [8.2 to 32.7]
  adjusted | 13.0 [4.0 to 34.6] | 17.0 [8.3 to 31.6]
Statistical Analysis 1: Comparison: Part 2, Placebo vs Part 2, BI 655064 120mg (RA); unadjusted; Test type: Superiority or Other; p = 0.3938, one-sided exact test (see description); one-sided exact test for superiority testing; risk difference, unadjusted = 4.5, 95% CI 2-sided [-18.4 to 22.3] — The exact 95% confidence interval was calculated by Clopper and Pearson
Statistical Analysis 2: Comparison: Part 2, Placebo vs Part 2, BI 655064 120mg (RA); adjusted; Test type: Superiority or Other; risk difference, adjusted = 4.0, 95% CI 2-sided [-18.9 to 21.1] — The 95 % confidence interval was determined by root method to determine the cumulative distribution function. Adjusted for treatment, region and anti-TNF history

8. Secondary Outcome: Part 2: EULAR Disease Activity Score in 28 Joints and C-reactive Protein (DAS28-CRP) at Week 12
Description: Assessed by European League Against Rheumatism (EULAR) categorization as good, moderate, or nonresponders based on improvement from baseline using the DAS28-CRP at week 12. In this outcome measure the frequency of EULAR response rates (change from the day of first dose to the day of visit 14 in week 12) are presented. DAS28-CRP is calculated as 0.56*√(TJC) + 0.28*√(SJC) + 0.36*Ln(CRP+1) + 0.014*VAS + 0.96. The total score ranges from 1.0 to 9.4, where a higher score indicates a better outcome.
  EULAR response states were classified as follows:
  good responders were patients with an improvement of >1.2 and a present score of ⩽3.2;
  moderate responders were patients with an improvement of >0.6 to ⩽1.2 and a present score of ⩽5.1, or an improvement of >1.2 and a present score of >3.2;
  non-responders were any patients with an improvement of ⩽0.6, or patients with an improvement of >0.6 to ⩽1.2 and a present score of >5.1.
  Improvement (impr.) is abbreviated in the category names.
Time Frame: baseline (day 1) and week 12 (day 85)
Population: FAS (observed cases)
Measure: Number; unit: Percentage of participants
Arm/Group | Part 2, Placebo | Part 2, BI 655064 120mg (RA)
Number analyzed (Participants) | 20 | 39
Percentage of participants
  DAS28-CRP <=3.2, improvement (>0.6 and <=1.2) | 5.0 | 2.6
  DAS28-CRP <=3.2, improvement <=0.6 | 0.0 | 0.0
  DAS28-CRP (>3.2 and <=5.1), improvement >1.2 | 25.0 | 35.9
  DAS28-CRP (>3.2 and <=5.1), impr. (>0.6 and <=1.2) | 5.0 | 7.7
  DAS28-CRP (>3.2 and <=5.1), improvement <=0.6 | 10.0 | 2.6
  DAS28-CRP >5.1, improvement >1.2 | 10.0 | 0.0
  DAS28-CRP>5.1, improvement (>0.6 and <=1.2) | 10.0 | 7.7
  DAS28-CRP >5.1, improvement <=0.6 | 10.0 | 7.7
  DAS28-CRP <=3.2, improvement >1.2 | 25.0 | 35.9

9. Secondary Outcome: Part 2: EULAR DAS28-ESR at Week 12
Description: Response as assessed by European League Against Rheumatism (EULAR) using Disease activity score in 28 joints and the erythrocyte sedimentation rate (DAS28-ESR) at week 12. In this outcome measure the frequency of EULAR response rates (change from the day of first dose to the day of visit 14 in week 12) are presented. DAS28-ESR is calculated as 0.56*√(TJC) + 0.28*√(SJC) + 0.70 *Ln(ESR) + 0.014*VAS. The total score ranges from 0 to 9.4, where a higher score indicates a better outcome.
  EULAR response states were classified as follows:
  good responders were patients with an improvement of >1.2 and a present score of ⩽3.2;
  moderate responders were patients with an improvement of >0.6 to ⩽1.2 and a present score of ⩽5.1, or an improvement of >1.2 and a present score of >3.2;
  non-responders were any patients with an improvement of ⩽0.6, or patients with an improvement of >0.6 to ⩽1.2 and a present score of >5.1.
  Improvement (impr.) is abbreviated in the category names.
Time Frame: baseline (day 1) and week 12 (day 85)
Population: FAS (observed cases)
Measure: Number; unit: Percentage of participants
Arm/Group | Part 2, Placebo | Part 2, BI 655064 120mg (RA)
Number analyzed (Participants) | 20 | 39
Percentage of participants
  DAS28-ESR <=3.2, improvement >1.2 | 10.5 | 20.5
  DAS28-ESR <=3.2, improvement (>0.6 and <=1.2) | 0.0 | 0.0
  DAS28-ESR <=3.2, improvement <=0.6 | 0.0 | 0.0
  DAS28-ESR (>3.2 and <=5.1), improvement >1.2 | 42.1 | 51.3
  DAS28-ESR (>3.2 and <=5.1), impr. (>0.6 and <=1.2) | 5.3 | 5.1
  DAS28-ESR (>3.2 and <=5.1), improvement <=0.6 | 0.0 | 0.0
  DAS28-ESR >5.1, improvement >1.2 | 21.1 | 10.3
  DAS28-ESR >5.1, improvement (>0.6 and <=1.2) | 5.3 | 7.7
  DAS28-ESR >5.1, improvement <=0.6 | 15.8 | 5.1

10. Secondary Outcome: Part 2: Percentage of Patients With a Decrease in DAS28-CRP of >1.2 at Week 12
Description: Percentage of patients who had a decrease of >1.2 on the Disease activity score in 28 joints and C-reactive protein (DAS28-CRP) at week 12 (day 85) compared to baseline. The adjusted absolute risk difference was adjusted for treatment, region and anti-TNF history. DAS28-CRP is calculated using Tender Joint Count 28 (TJC28), Swollen Joint Count 28 (SJC28), C-reactive protein (CRP) (in mg/L), Patient's Global Assessment of Arthritis Disease Activity (PtGA) (visual analogue scale with values from 0=best to 100=worst), where the total score is calculated as follows: 0.56*√(TJC) + 0.28*√(SJC) + 0.36*Ln(CRP+1) + 0.014*VAS + 0.96. The total score ranges from 1.0 to 9.4, where a higher score indicates a better outcome.
Time Frame: baseline (day 1) and week 12 (day 85)
Population: FAS (Last observation carried forward)
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part 2, Placebo | Part 2, BI 655064 120mg (RA)
Number analyzed (Participants) | 22 | 44
Percentage of participants
  Unadjusted | 59.1 [36.4 to 79.3] | 65.9 [50.1 to 79.5]
  Adjusted | 58.2 [36.7 to 77.0] | 67.1 [51.6 to 79.6]
Statistical Analysis 1: Comparison: Part 2, Placebo vs Part 2, BI 655064 120mg (RA); unadjusted; Test type: Superiority or Other; Risk difference = 6.8, 95% CI 2-sided [-17.6 to 32.7] — The exact 95% confidence interval was calculated by Clopper and Pearson
Statistical Analysis 2: Comparison: Part 2, Placebo vs Part 2, BI 655064 120mg (RA); adjusted; Test type: Superiority or Other; risk difference, adjusted = 8.9, 95% CI 2-sided [-15.9 to 34.2] — [estimate comment as in outcome 7, analysis 2]

11. Secondary Outcome: Part 2: Change in DAS28-CRP Score at Week 12
Description: Change at week 12 in the Disease activity score in 28 joints and C-reactive protein (DAS28-CRP) compared with the score at baseline. The mean was adjusted for region, anti-TNF history and baseline DAS28-CRP. DAS28-CRP is calculated using Tender Joint Count 28 (TJC28), Swollen Joint Count 28 (SJC28), C-reactive protein (CRP) (in mg/L), Patient's Global Assessment of Arthritis Disease Activity (PtGA) (visual analogue scale with values from 0=best to 100=worst), where the total score is calculated as follows: 0.56*√(TJC) + 0.28*√(SJC) + 0.36*Ln(CRP+1) + 0.014*VAS + 0.96. The total score ranges from 1.0 to 9.4, where a higher score indicates a better outcome.
Time Frame: baseline (day 1) and week 12 (day 85)
Population: FAS (last observation carried forward)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Part 2, Placebo | Part 2, BI 655064 120mg (RA)
Number analyzed (Participants) | 22 | 44
units on a scale
  Mean | -1.45 (0.238) | -1.61 (0.140)
  Adjusted mean | -1.47 (0.215) | -1.60 (0.151)
Statistical Analysis 1: Comparison: Part 2, Placebo vs Part 2, BI 655064 120mg (RA); difference calculated as BI 655064 120mg minus placebo; Test type: Superiority or Other; Adjusted mean = -0.14, 95% CI 2-sided [-0.67 to 0.39], Standard Error of Mean 0.266 — difference calculated as BI 655064 120mg minus placebo. The ANCOVA model was used. In this model the mean was adjusted for region, anti-TNF history and baseline DAS28-CRP

ADVERSE EVENTS:
Time Frame: from first administration of study medication (day 1) up to day 64 (dosing groups 80, 120, 180mg) or up to day 78 post-treatment (dosing group 240mg) in part 1 and up to 141 days in part 2.
Description: Treated set (TS): This patient set includes all subjects who were dispensed study medication and were documented to have taken at least one dose of investigational treatment.
Groups:
- Part 1, BI 655064 80mg (HV): Part 1, HV: 80 mg of BI 655064 injected subcutaneous on days 1, 8, 15, and 22 (once weekly, for 4 weeks) followed by 6 weeks follow-up period.
- Part 1, BI 655064 120mg (HV): Part 1, HV: 120 mg of BI 655064 injected subcutaneous on days 1, 8, 15, and 22 (once weekly, for 4 weeks) followed by 6 weeks follow-up period.
- Part 1, BI 655064 180mg (HV): Part 1, HV: 180 mg of BI 655064 injected subcutaneous on days 1, 8, 15, and 22 (once weekly, for 4 weeks) followed by 6 weeks follow-up period.
- Part 1, BI 655064 240mg (HV): Part 1, HV: 240mg of BI 655064 injected subcutaneous on days 1, 8, 15, and 22 (once weekly, for 4 weeks) followed by 8 weeks follow-up period.
- Part 1, Placebo (HV): Part 1, HV: Placebo injected subcutaneous on days 1, 8, 15, and 22 (once weekly, for 4 weeks) followed by 6 weeks (80, 120, and 180mg dosing group) or 8 weeks (240mg dosing group) follow-up period.
Arm/Group | Part 1, BI 655064 80mg (HV) | Part 1, BI 655064 120mg (HV) | Part 1, BI 655064 180mg (HV) | Part 1, BI 655064 240mg (HV) | Part 1, Placebo (HV) | Part 2, BI 655064 120mg (RA) | Part 2, Placebo BI 655064 120mg (RA)
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 2/44 | 2/23
Other Adverse Events (participants affected / at risk) | 7/8 | 6/8 | 6/8 | 6/8 | 7/8 | 29/44 | 17/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1, BI 655064 80mg (HV) (N=8) | Part 1, BI 655064 120mg (HV) (N=8) | Part 1, BI 655064 180mg (HV) (N=8) | Part 1, BI 655064 240mg (HV) (N=8) | Part 1, Placebo (HV) (N=8) | Part 2, BI 655064 120mg (RA) (N=44) | Part 2, Placebo BI 655064 120mg (RA) (N=23)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cardiopulmonary failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1, BI 655064 80mg (HV) (N=8) | Part 1, BI 655064 120mg (HV) (N=8) | Part 1, BI 655064 180mg (HV) (N=8) | Part 1, BI 655064 240mg (HV) (N=8) | Part 1, Placebo (HV) (N=8) | Part 2, BI 655064 120mg (RA) (N=44) | Part 2, Placebo BI 655064 120mg (RA) (N=23)
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Eye pain (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Photophobia (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0
Food poisoning (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 1
Toothache (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Catheter site oedema (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 1 | 1 | 1 | 0 | 2
Injection site bruising (General disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Injection site pain (General disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 0
Injection site rash (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Vessel puncture site bruise (General disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Liver disorder (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 2
Chlamydial infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fungal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 1 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 6 | 5
Pharyngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Rhinitis (Infections and infestations) | 0 | 1 | 2 | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 2 | 2 | 1 | 1 | 1 | 1
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 | 1
Viral infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 3 | 2 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 2 | 1 | 0 | 0 | 1 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sunburn (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 2
Joint laxity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 3 | 2 | 3 | 1 | 4 | 3 | 3
Lethargy (Nervous system disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Dyspareunia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 2 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0 | 1 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Xeroderma (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.